CLINICAL TRIAL: NCT04653415
Title: The Impact of Pre-emptive Large Doses of Methylprednisolone Combined With Gabapentin on Pain Treatment and Convalescence After Total Knee Arthroplasty in Elderly: A Double-blind Randomized Study
Brief Title: Large Doses of Methylprednisolone Combined With Gabapentin in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Henryk Liszka, Principial Investigator, Assisstant Professor, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1072.6120.11.2020
Record Dates: First submitted 2020-11-21; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Arthroplasty Complications; Knee Osteoarthritis; Pain, Postoperative; Perioperative Complication
Keywords: total knee arthroplasty; pre-emptive analgesia; methylprednisolone; gabapentin; opioid dose; pain intensity; infection rate
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative; Pain | interventions — Gabapentin; Methylprednisolone; Tablets; Saline Solution; Injections

STUDY DESIGN:
Intervention Model Description: two groups: the study and controls
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants of the study are blinded to receive methylprednisolone with gabapentin (the study group) or placebo (the controls group). Only nurse knows if administer drug or placebo. Both outcome assessor and investigator are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): The study group will receive as "pre-emptive" analgesia a single dose of 300 mg oral gabapentin and 125 mg intravenous methylprednisolone.
  Interventions: Drug: Gabapentin 300mg; Drug: Methylprednisolone 125 mg
- Controls group (Placebo Comparator): The controls group will receive placebo orally - a tablet without any pharmacological properties, intravenously - saline solution.
  Interventions: Drug: Tablet; Drug: Normal Saline 10 mL Injection

INTERVENTIONS:
Drug: Gabapentin 300mg — The study group will receive as "pre-emptive" analgesia a single dose of 300 mg oral gabapentin and 125 mg intravenous methylprednisolone.
  Arms: Study Group
Drug: Methylprednisolone 125 mg — The study group will receive as "pre-emptive" analgesia a single dose of 300 mg oral gabapentin and 125 mg intravenous methylprednisolone.
  Arms: Study Group
Drug: Tablet — The controls group will receive placebo orally - a tablet without any pharmacological properties, intravenously - normal saline solution
  Arms: Controls group
Drug: Normal Saline 10 mL Injection — The controls group will receive placebo orally - a tablet without any pharmacological properties, intravenously - normal saline solution
  Arms: Controls group

SUMMARY:
The aim of the study was to assess whether administration of gabapentin and methylprednisolone as "pre-emptive analgesia" in a group of patients above 65 years of age would be effective in complex pain management therapy following total knee arthroplasty (TKA). For the study investigators will qualify one hundred seventy, above 65 years old patients. The participants will be double-blind randomized into two groups: the study and controls The study group will receive as "pre-emptive" analgesia a single dose of 300 mg oral gabapentin and 125 mg intravenous methylprednisolone, while the others placebo. Perioperatively, all the patients will receive opioid and nonopioid analgesic agents calculated for 1 kg of body weight. Investigators will measure the levels of inflammatory markers (leukocytosis, C-reactive protein - CRP), pain intensity level at rest (numerical rating scale - NRS), the life parameters and all complications.

DETAILED DESCRIPTION:
The aim of the study was to assess whether administration of gabapentin and methylprednisolone as "pre-emptive analgesia" in a group of patients above 65 years of age would be effective in complex pain management therapy following total knee arthroplasty (TKA).170 patients operated on due to unilateral TKA will be double-blinded randomized into two groups: the study and the controls. Exclusion criteria are: clinical situation that 1/ restricted glucocorticoid administration: diabetes type 1 and 2, CRP levels above normal values (≥5 mg/l), chronic steroid treatment, peptic ulcers treated in the past 30 days and 2/and the chronic pain in the course of gonarthrosis, high intensity requiring use opioids.

The participants of the study will be subjected to the standardized procedure of subarachnoid anesthesia with subsequent unilateral femoral nerve block at the operated side, followed by the surgical procedure - unilateral TKA. The study group will receive as "pre-emptive" analgesia a single dose of 300 mg oral gabapentin and 125 mg intravenous methylprednisolone, while the others placebo. Prior to anesthesia induction, the patients receive: anti-infection prophylactics intravenous cephazolin 2.0 g, for hemostasis control - tranexamic acid 1.0 g, an anti-emetic agent - ondansetron 8 mg. Fluid supply (crystalloids) will be standardized: 12 ml/kg in the first hour of surgery and 6 ml/kg in the following hours, packed red blood cells if blood loss exceeded 600 ml and hemoglobin concentration <10g/l during the time of operation. Pain management will be carried out based on the results of the NRS scales at rest. Every 6 hours NRS will be checked and intravenous PCA (patient-controlled analgesia) oxycodone hydrochloride, if pain was ≥4 points NRS or intravenous paracetamol, metamizole, if the pain was 2 - 4 NRS points will be administered, all pain medications will be calculated for 1 kg of body weight. In keeping with the ERAS (Enhanced Recovery After Surgery) protocol, on the day of surgery the patients will receive orally fluids and meals, will be mobilized and rehabilitated.

The study was approved by the institutional review board (nr 1072.6120.11.2020). Oral and written informed consent to participate in the study will be collected from all participants of the study. The statistical analysis of the groups will be performed to asess the demographic dates, life parameters, general condition in keeping with the ASA (American Society of Anesthesiology), POSSUM (Physiologic and Operative Severity Score for the enUmeration of Mortality and Morbidity) score, total dose of analgesic medications administered parenterally calculated for 1 kg of body mass in response to value of NRS at rest on day 0, time of administration the first dose, and duration of peripheral nerve block. On the day of surgery and on subsequent days, determinations will be made of glycemia levels and inflammatory markers: C-reactive protein (CRP) and leukocytosis levels.

ELIGIBILITY:
Inclusion Criteria:

* patients over 65 years old operated on unilateral total knee arthroplasty

Exclusion Criteria:

* diabetes type 1 and 2,
* CRP levels above normal values (≥5 mg/l),
* chronic steroid treatment,
* peptic ulcers treated in the past 30 days,
* chronic pain in the course of gonarthrosis,

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity assessed by NRS | change in every 6 hours on day 0
  The level of postoperative pain measured in the numerical rating scale (NRS) at rest (minimum 0 - no pain, maximum 10 - the maximum of pain).
the dose of parenteral analgesics agents | 24 hours
  Dose of oxycodone hydrochloride in mg/kg body weight, paracetamol in mg/kg body weight, metamizole in g/kg body weight
C-reactive protein (CRP) level | change in 0,1,2,3 days after surgery
  C-reactive protein (CRP) level measured in mg/l
Leukocytosis level | change in 0,1,2,3 days after surgery
  Leukocytosis level measured in µL
Adverse effects | 0 day after surgery
  The occurrence of adverse effects that would delay early rehabilitation, possible complication development, perioperative mortality to the POSSUM scale, comorbidities
Adverse effects | 1 day after surgery
  The occurrence of adverse effects that would delay early rehabilitation, possible complication development, perioperative mortality to the POSSUM scale, comorbidities
Adverse effects | 2 day after surgery
  The occurrence of adverse effects that would delay early rehabilitation, possible complication development, perioperative mortality to the POSSUM scale, comorbidities
Adverse effects | 3 day after surgery
  The occurrence of adverse effects that would delay early rehabilitation, possible complication development, perioperative mortality to the POSSUM scale, comorbidities
Adverse effects | 14 day after surgery
  The occurrence of adverse effects that would delay early rehabilitation, possible complication development, perioperative mortality to the POSSUM scale, comorbidities

SECONDARY OUTCOMES:
Duration of femoral nerve blockade | on the day of surgery
  The time of femoral nerve block
Blood glucose level | change in 0,1,2,3 days after surgery
  The level of glucose in blood in mmol/l

OTHER OUTCOMES:
Mean age | the day of surgery
  Mean age in years
Mean hospitalization time | from admission to hospital till 14 days after surgery
  Mean hospitalization time in days
Mean postoperative hospitalization time | change from 0 till 14 days after surgery
  Mean postoperative hospitalization time in days
Postoperative Mean Arterial Pressure (MAP) | change in 0,1,2,3 days after surgery
  Postoperative Mean Arterial Pressure (MAP) measured in mmHg
Postoperative pulse | change in 0,1,2,3 days after surgery
  Postoperative pulse (x/min)) measured in x/min
Postoperative saturation (Sp02) of the arterial blood | change in 0,1,2,3 days after surgery
  Postoperative saturation (Sp02) of the arterial blood measured in %
Physiological and Operative Severity Score for the enUmeration of Mortality and morbidity (POSSUM) morbidity | the day of the surgery
  Physiological and Operative Severity Score for the enUmeration of Mortality and morbidity (POSSUM) morbidity measured in %
Physiological and Operative Severity Score for the enUmeration of Mortality and morbidity (POSSUM) mortality | the day of the surgery
  Physiological and Operative Severity Score for the enUmeration of Mortality and morbidity (POSSUM) mortality measured in %
Physiological and Operative Severity Score for the enUmeration of Mortality and morbidity (POSSUM) physiological score | the day of the surgery
  Physiological and Operative Severity Score for the enUmeration of Mortality and morbidity (POSSUM) physiological score measured in points (minimum 12, maximum 96)
American Society of Anesthesiology Score (ASA) | the day of the surgery
  American Society of Anesthesiology Score (ASA), grade I-IV

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital in Krakow, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Lamplot JD, Wagner ER, Manning DW. Multimodal pain management in total knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Feb;29(2):329-34. doi: 10.1016/j.arth.2013.06.005. Epub 2013 Jul 11. PMID 23850410
- [Background] Kehlet H, Lindberg-Larsen V. High-dose glucocorticoid before hip and knee arthroplasty: To use or not to use-that's the question. Acta Orthop. 2018 Oct;89(5):477-479. doi: 10.1080/17453674.2018.1475177. Epub 2018 May 21. No abstract available. PMID 29781366
- [Background] Luna IE, Kehlet H, Petersen MA, Aasvang EK. Clinical, nociceptive and psychological profiling to predict acute pain after total knee arthroplasty. Acta Anaesthesiol Scand. 2017 Jul;61(6):676-687. doi: 10.1111/aas.12899. Epub 2017 May 16. PMID 28508511
- [Background] Jorgensen CC, Pitter FT, Kehlet H; Lundbeck Foundation Center for Fast-track Hip and Knee Replacement Collaborative Group. Safety aspects of preoperative high-dose glucocorticoid in primary total knee replacement. Br J Anaesth. 2017 Aug 1;119(2):267-275. doi: 10.1093/bja/aex190. PMID 28854533
- [Background] Hartman J, Khanna V, Habib A, Farrokhyar F, Memon M, Adili A. Perioperative systemic glucocorticoids in total hip and knee arthroplasty: A systematic review of outcomes. J Orthop. 2017 Apr 12;14(2):294-301. doi: 10.1016/j.jor.2017.03.012. eCollection 2017 Jun. PMID 28442852
- [Background] Lindberg-Larsen V, Ostrowski SR, Lindberg-Larsen M, Rovsing ML, Johansson PI, Kehlet H. The effect of pre-operative methylprednisolone on early endothelial damage after total knee arthroplasty: a randomised, double-blind, placebo-controlled trial. Anaesthesia. 2017 Oct;72(10):1217-1224. doi: 10.1111/anae.13983. Epub 2017 Jul 26. PMID 28744857
- [Background] Gadek A, Liszka H, Zajac M. The effect of pre-operative high doses of methylprednisolone on pain management and convalescence after total hip replacement in elderly: a double-blind randomized study. Int Orthop. 2021 Apr;45(4):857-863. doi: 10.1007/s00264-020-04802-8. Epub 2020 Sep 17. PMID 32940751
- [Background] Lee JK, Chung KS, Choi CH. The effect of a single dose of preemptive pregabalin administered with COX-2 inhibitor: a trial in total knee arthroplasty. J Arthroplasty. 2015 Jan;30(1):38-42. doi: 10.1016/j.arth.2014.04.004. Epub 2014 Apr 13. PMID 24851793
- [Background] Lubis AMT, Rawung RBV, Tantri AR. Preemptive Analgesia in Total Knee Arthroplasty: Comparing the Effects of Single Dose Combining Celecoxib with Pregabalin and Repetition Dose Combining Celecoxib with Pregabalin: Double-Blind Controlled Clinical Trial. Pain Res Treat. 2018 Aug 7;2018:3807217. doi: 10.1155/2018/3807217. eCollection 2018. PMID 30174951
- [Background] Osinski T, Bekka S, Regnaux JP, Fletcher D, Martinez V. Functional recovery after knee arthroplasty with regional analgesia: A systematic review and meta-analysis of randomised controlled trials. Eur J Anaesthesiol. 2019 Jun;36(6):418-426. doi: 10.1097/EJA.0000000000000983. PMID 30950899
- [Background] Berg U, BuLow E, Sundberg M, Rolfson O. No increase in readmissions or adverse events after implementation of fast-track program in total hip and knee replacement at 8 Swedish hospitals: An observational before-and-after study of 14,148 total joint replacements 2011-2015. Acta Orthop. 2018 Oct;89(5):522-527. doi: 10.1080/17453674.2018.1492507. Epub 2018 Jul 9. PMID 29985681
- [Background] Pamilo KJ, Torkki P, Peltola M, Pesola M, Remes V, Paloneva J. Fast-tracking for total knee replacement reduces use of institutional care without compromising quality. Acta Orthop. 2018 Apr;89(2):184-189. doi: 10.1080/17453674.2017.1399643. Epub 2017 Nov 21. PMID 29160123
- [Background] Shen S, Gao Z, Liu J. The efficacy and safety of methylprednisolone for pain control after total knee arthroplasty: A meta-analysis of randomized controlled trials. Int J Surg. 2018 Sep;57:91-100. doi: 10.1016/j.ijsu.2018.07.009. Epub 2018 Aug 16. PMID 30120990
- [Background] Lei Y, Xie J, Xu B, Xie X, Huang Q, Pei F. The efficacy and safety of multiple-dose intravenous tranexamic acid on blood loss following total knee arthroplasty: a randomized controlled trial. Int Orthop. 2017 Oct;41(10):2053-2059. doi: 10.1007/s00264-017-3519-x. Epub 2017 May 31. PMID 28567578